CLINICAL TRIAL: NCT05933863
Title: Molecular Subtyping of Extensive Stage Small Cell Lung Cancer and Relevent Clinical Significance
Acronym: MOSAIC
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2021YJZ97
Record Dates: First submitted 2023-06-24; First posted 2023-07-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: SCLC,Extensive Stage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immunotherapy cohort: Extensive stage SCLC patients receiving first-line chemotherapy plus PD-(L)1 antibody treatment will be enrolled in this cohort. Baseline tumor tissue samples and peripheral blood samples will be collected for transcriptome and immunohistochemistry analysis etc.
  Interventions: Drug: PD-(L)1 antibody immunotherapy
- chemotherapy cohort: Extensive stage SCLC patients receiving only first-line etoposide plus platinum chemotherapy will be enrolled in this cohort. Baseline tumor tissue samples and peripheral blood samples will be collected for transcriptome and immunohistochemistry analysis etc.

INTERVENTIONS:
Drug: PD-(L)1 antibody immunotherapy — The treatment regimen involved in this study follows guidelines for the first-line treatment of extensive stage SCLC: cisplatin+etoposide or carboplatin+etoposide and PD-(L)1 inhibitor.
  Groups: immunotherapy cohort

SUMMARY:
To validate the predictive value of transcriptome-based molecular subtyping of extensive stage small cell lung cancer (SCLC) for the efficacy of programmed death-1(PD-1)/programmed death-ligand1(PD-L1) inhibitor in the first line setting; to explore the differences of immune microenvironment between different SCLC subtypes to reveal the mechanisms of immunotherapy resistance of SCLC

DETAILED DESCRIPTION:
This retrospective observational study examines the predictive value of transcriptome-based molecular subtyping of extensive stage SCLC for PD-1/PD-L1 inhibitor efficacy and explores immune microenvironment differences between subtypes to uncover immunotherapy resistance mechanisms. Patients with extensive stage SCLC receiving first-line standard treatment are enrolled, and baseline tumor tissue and peripheral blood samples are collected for transcriptome sequencing and immunohistochemistry (IHC). Based on results, patients are classified into four molecular subtypes, and treatment efficacy and safety are recorded. The study compares the efficacy between SCLC subtypes to determine if molecular typing predicts immunotherapy efficacy and investigates immune microenvironment differences between subtypes to uncover resistance mechanisms. Treatment regimens follow first-line extensive stage SCLC guidelines, including cisplatin+etoposide or carboplatin+etoposide and PD-(L)1 inhibitors, with options determined by the supervising physician.

ELIGIBILITY:
Inclusion Criteria:

* The enrolled subjects shall meet all the following conditions at the same time.

  1. Male or female, aged 18 to 100 years
  2. Patients with untreated advanced small cell lung cancer clearly diagnosed by histopathology
  3. Be able to provide tumor biopsy tissue sample for molecular analysis
  4. Eastern Cooperative oncology Group (ECOG) score: 0~2
  5. Expected survival of more than 3 months.
  6. Has at least 1 measurable or evaluable tumor lesion with a longest diameter ≥ 10 mm at baseline (in case of lymph nodes, a shortest diameter ≥ 15 mm is required) according to RECIST v1.1
  7. Received first-line chemotherapy or chemotherapy＋PD-(L)1 inhibitor and be able to provide complete treatment information and efficacy evaluation results.
  8. Voluntary signed informed consent and expected good compliance.

Exclusion Criteria:

* Those meeting any of the following conditions may not be included.

  1. Patient unable to tolerate chemotherapy.
  2. Patients unable to provide tumor tissue samples for testing
  3. Patients with other malignant tumors or a history of other malignant tumors
  4. Patients have any other reason to be unfit to participate in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adults (18-100 years) with untreated advanced SCLC. Eligible patients have an ECOG score of 0~2, an expected survival >3 months, and can provide tumor biopsy samples for transcripsome testing. They must have received first-line chemotherapy or chemotherapy combined with a PD-L1 inhibitor.
  Participants are divided into two arms: Chemotherapy (80-100 cases) and Immunotherapy+chemotherapy (80-100 cases). Exclusion criteria include intolerance to chemotherapy, inability to provide tumor tissue samples, presence/history of other malignant tumors, and other reasons deeming them unfit for the study.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2022.4.1-2023.12.31
  From the start of first-line treatment until disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | 2022.4.10-2024.12.31
  From the start of first-line treatment until death due to any cause
Objective response rate | 2022.4.10-2023.12.31
  The tumor size was calculated by computed tomography or magnetic resonance Imaging scan, the best response was evaluated based on Response Evaluation Criteria in Solid Tumors (RECISTVersion1.1)
molecular subtyping and tumor microenvironment biomarkers | 2022.4.10-2023.12.31
  The molecular subtyping was carried out based on transcripsome sequencing following the method in published article PMID: 33482121, the tumor microenvironment biomarkers include tumor infiltrated immune cells and specific gene expression evaluated by transcripsome and Multiplex immunohistochemical analysis etc.

CONTACTS AND LOCATIONS:
Overall Officials: Minglei Zhuo, Physician, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT05933863/Prot_SAP_000.pdf